CLINICAL TRIAL: NCT03926585
Title: Longtime Effect of Combination Treatment With L-thyroxine (L-T4) and Liothyronine (L-T3) in Patients With Persistent Hypothyroid Symptoms - Relation to Polymorphisms (SNP) in the DIO2 and the MCT10 Gene
Brief Title: Variations in the DIO2 and MCT10 Genes and Effect of Triiodothyronine Treatment
Status: Completed | Type: Observational
Sponsor: Birte Nygaard (Other)
Responsible Party: Sponsor-Investigator, Birte Nygaard, Chief Physician, Ph.D, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: T3SNP
Record Dates: First submitted 2019-04-15; First posted 2019-04-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Patients in combination therapy due to persistent symptoms on L-thyroxin mono-therapy who experience a longtime effect of triiodothyronine treatment.
- Non-responders: Patients who have tried combination therapy due to persistent symptoms on L-thyroxin mono-therapy, but did not experience a longtime effect.

SUMMARY:
Hypothesis: Variations in the deiodinase 2 gene and monocarboxylate transporter 10 gene is associated with improvement in quality of life after initiation of combination therapy with L-Thyroxine and Liothyronine in patients with persistent hypothyroid symptoms despite conventional L-thyroxine mono-therapy.

Purpose: To re-test this hypothesis in patients with continued perceived effect of Liothyronine treatment at least one year after initiation in a patient population more representing of daily clinical practice. The study will help determine whether testing of specific gene variations might predict longtime effect of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the department of endocrinology with the diagnose hypothyroidism because of persistent hypothyroid symptoms despite treatment with L-thyroxine mono-therapy and normal and stable TSH (for at least 6 months).
* Started in combination therapy with L-thyroxine and Liothyronine in an approximately 17/1 ratio
* Exclusion of an alternative explanation for persistent hypothyroid symptoms

Exclusion Criteria:

* Initiation of L-thyroxine treatment in patients with s-TSH below upper normal limit (with assay in current use, that is TSH < 4 mU/L)
* Ongoing pregnancy
* Age below 18 years or above 80 years.
* Patients who do not read and understand information material given
* Patients who are not competent to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in this study have been diagnosed with hypothyroidism and have had persistent hypothyroid symptoms despite L-thyroxine mono-therapy. They have all been referred to the department of endocrinology and have been examined by a trained endocrinologist. All patients have at least one year before the study initiated combination therapy with L-thyroxine and Liothyronine.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Polymorphisms in DIO2/MCT10 and triiodothyronine treatment | Single assessment point, from 1-10 years after initiation of combination therapy
  Group 1(responders) and group 2(non-responders) are compared with regard to polymorphisms in the DIO2 gene and the MCT10 gene. Polymorphisms will be determined from DNA in a blood sample

SECONDARY OUTCOMES:
Proportion treated with triiodothyronine | Single assessment point, from 1-10 years after initiation of combination therapy
  How many patients are treated with triiodothyronine at least one year after initiation of combination therapy.
Quality of life questionnaire | Single assessment point, from 1-10 years after initiation of combination therapy
  Patients are scored on the ThyPRO questionnaire and a hypothyroid symptoms questionnaire.
Who controls the treatment? | Single assessment point, from 1-10 years after initiation of combination therapy
  Patients report whether treatment is controlled by 1) a general practitioner 2) Patient self 3) other type of healthcare professional 4) a certified endocrinologist or 5) other
How is current treatment controlled? | Single assessment point, from 1-10 years after initiation of combination therapy
  Patients report if current treatment is for example controlled by using blood samples or only on the basis of symptoms.
Have therapy changed after the patient left the department of endocrinology? | Single assessment point, from 1-10 years after initiation of combination therapy
  Current hypothyroidism treatment and doses of medication
TSH | Single assessment point, from 1-10 years after initiation of combination therapy
  Is the patient well regulated? Normal TSH: 0.1-4.0 (depending on assay used). Over-treatment: TSH < 0.1 (depending on assay used). Under-treatment: TSH>4 (depending on assay used).
Osteoporosis | Single assessment point, from 1-10 years after initiation of combination therapy
  DXA-scan
Risk of arrhythmia | Single assessment point, from 1-10 years after initiation of combination therapy
  Puls and blood pressure is measured. If arrhythmia is suspected, an ECG is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Birte Nygaard, Ph.D., Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided